CLINICAL TRIAL: NCT04512729
Title: Detection Of Colonic Polyps In India: Diagnostic Colonoscopy
Acronym: DoCPI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Principal Investigator, Asian Institute of Gastroenterology, India
Other Study IDs: DoCPI
Record Dates: First submitted 2020-08-12; First posted 2020-08-13 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Colonic Polyp; Colonic Adenoma; Colonic Neoplasms
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Colonoscopy — For all patients, either moderate sedation with intravenous midazolam or conscious sedation with intravenous propofol will be administered in a standard fashion prior to undergoing colonoscopy.
  The colonoscope will be inserted and cecum will be intubated. Photo documentation of the cecum will be performed. The colonic mucosa will be carefully visualized upon withdrawal of the colonoscope.
  The time spent in inspecting the mucosa during withdrawal of the colonoscope will be documented as the "withdrawal time". Meticulous technique will be employed during the withdrawal phase with special efforts to visualize portions of colonic mucosa on the proximal aspects of haustral folds, flexures and valves.All polyps detected will be documented: size, location, and morphology. Photo documentation of the polyps will be performed.

SUMMARY:
Colorectal carcinoma (CRC) is the third most common cancer in male and female worldwide. In India, it is the fourth most common cause of cancer in males and third most common cancer in female. Age, smoking, colonic adenomatous polyp, family history are traditional risk factor for CRC. The vast majority of CRC results from malignant transformation from adenoma, which is called as adenoma carcinoma sequence. These adenomatous polyps grows slowly over many years and malignant transformation eventually occurs over 10 years. So, the early detection and removal of polyp at early stage should benefit in preventing CRC.

DETAILED DESCRIPTION:
The third most common cancer in both male and female is colorectal carcinoma (CRC) worldwide. In India, it is the fourth most common cause of cancer in males and third most common cancer in females. The age - standardized rates of CRC in India have been estimated to be 4.2 and 3.2/100000 for males and females, respectively. Age, smoking and colonic adenoma along with family history is considered as traditional risk factors for CRC. The US National Polyp study demonstrated that colonoscopy and polypectomy could prevent 76% to 90% of colorectal cancers. The vast majority of CRC result from malignant transformation from adenomas. This is called adenoma - carcinoma sequence, these adenomatous polyps grows slowly over many years and malignant transformation eventually occurs. The time span for this transformation is on an average 10 years. So, the detection and removal of polyp at early stage on adenoma - carcinoma sequence should benefit in preventing CRC.

The prevalence of adenoma, utilization of colonoscopy for its detection and subsequent reduction in CRC has been well studied and established in western population. This has led to formulation of national screening colonoscopy programs elsewhere. However, data from Indian subcontinent is scanty. In current study, at a large tertiary care center, we aimed to study prevalence of colonic polyps and adenoma who are undergoing diagnostic colonoscopy using high definition colonoscopy and characterizing with Narrow Band Imaging and to find associated demographic, social, personal and family related risk factors in patients with adenomas.

Methodology:

This will be a prospective, single center, observational study. All subjects referred for diagnostic colonoscopy will be prospectively enrolled.

Enrollment:

All subjects referred for the diagnostic colonoscopy will be enrolled. A member of the research team will approach each subject to discuss participation in the study, including background of the proposed study, inclusion and exclusion criteria, benefits and risks of the procedures and follow-up. If this is of interest to the subject, the informed consent form is discussed and presented. The subject must sign the consent form prior to enrollment. This form will have prior approval of the study site's Institutional Review Board (IRB). Failure to obtain informed consent renders the subject ineligible for the study.

Study equipment

Colonoscope:

Olympus HDWL colonoscope will be used to perform colonoscopies. Technical specifications include outer diameter 13.2 mm, instrument channel diameter 3.7 mm, air-water suction channels, field of view 170 degrees, 4-way angulations (180 degrees up and 180 degrees down, 160 degrees right and left), working length, 168 cm.

Colonoscopy procedure and definitions

For all patients, either moderate sedation with intravenous midazolam or conscious sedation with intravenous propofol will be administered in a standard fashion prior to undergoing colonoscopy.

The colonoscope will be inserted and cecum will be intubated. Photo documentation of the cecum will be performed. The colonic mucosa will be carefully visualized upon withdrawal of the colonoscope.

The time from the point of insertion of the colonoscope into the rectum to the intubation of cecum will be recorded with a stop watch by a research coordinator and will be documented as the "insertion time".

The time spent in inspecting the mucosa during withdrawal of the colonoscope will be documented as the "withdrawal time". During withdrawal of the colonoscope the stop watch will be stopped whenever mucosa is being cleaned, fluid/solid debris is suctioned or a polyp is being removed to ensure that the withdrawal time is the actual representation of the mucosal inspection time. Meticulous technique will be employed during the withdrawal phase with special efforts to visualize portions of colonic mucosa on the proximal aspects of haustral folds, flexures and valves.

All polyps detected will be documented: size, location, and morphology (using the Paris classification - Appendix A and Narrow Band Imaging classification - NICE and JNET). Photo documentation of the polyps will be performed.

Polyps will then be removed with a biopsy forceps or snare and sent for histopathological evaluation, each in a separate jar and labeled accordingly.

The bowel preparation will be evaluated and graded according to previously reported criteria using the Boston Bowel Preparation Scale. Complications including post colonoscopy pain, perforation or gastrointestinal bleeding (requiring intervention) will be recorded.

Adverse events:

The primary investigator at each site will monitor any adverse events reported to the study staff and determine if it's related to the study procedures including standard colonoscopy at the respective site. All adverse events will be monitored until a satisfactory resolution and will be reported to the local IRB within 5 days of knowledge. A table will be maintained for the adverse events in each arm and in case of any statistically significant adverse even rate in any arm, the primary investigator will make the decision to remove the treatment arm or stop the study. Because the risks of this proposed study are low, this program will not require a Data Safety and Monitoring Board. Instead, the Principal Investigator and clinical Site Investigators performing the endoscopies will be responsible for implementing a detailed Data and Safety Monitoring plan in compliance with the IRB guidelines.

Data integrity and safety:

All paper charts pertaining to the patient will be kept under lock and key in coordinators office away from the endoscopy area. The data will be entered in to a data base weekly after collection of histology reports. The data is password protected and stored on the AIG internal server where it will remain throughout the study. Computers and/or files will be password-protected. Only approved personnel by the IRB will have access to the file storage.

To protect subject confidentiality, each subject will be assigned a case study number. The subject's name is not to appear anywhere on the Case Report Forms (CRF's) or supporting documentation. A study log with the identifiable information will be kept in a separate folder to enable the investigators to assist in any research audit. No procedural data except the date of examination will be entered in to this log.

ELIGIBILITY:
Inclusion Criteria:

* Referral for diagnostic colonoscopy
* Ability to provide informed consent

Exclusion Criteria:

• Inability or not willing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects referred for the diagnostic colonoscopy will be enrolled. A member of the research team will approach each subject to discuss participation in the study, including background of the proposed study, inclusion and exclusion criteria, benefits and risks of the procedures and follow-up. If this is of interest to the subject, the informed consent form is discussed and presented. The subject must sign the consent form prior to enrollment. This form will have prior approval of the study site's Institutional Review Board (IRB). Failure to obtain informed consent renders the subject ineligible for the study
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Colonic Adenoma | 1 year
  To evaluate prevalence of colonic polyps and adenomas in Indian Population

SECONDARY OUTCOMES:
Risk factors for Colonic adenoma | 1 year
  1. To find possible risk factors associated with colonic adenoma to plan CRC screening program

CONTACTS AND LOCATIONS:
Locations (1):
- D Nageshwar Reddy, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers.

REFERENCES:
- [Derived] Jagtap N, Kalapala R, Rughwani H, Singh AP, Inavolu P, Ramchandani M, Lakhtakia S, Manohar Reddy P, Sekaran A, Tandan M, Nabi Z, Basha J, Gupta R, Memon SF, Venkat Rao G, Sharma P, Nageshwar Reddy D. Application of machine-learning model to optimize colonic adenoma detection in India. Indian J Gastroenterol. 2024 Oct;43(5):995-1001. doi: 10.1007/s12664-024-01530-4. Epub 2024 May 17. PMID 38758433